CLINICAL TRIAL: NCT04790799
Title: Occupational Hand Eczema - Establishment and Testing of a Prevention-concept With Focus on the Young Workforce
Brief Title: Occupational Hand Eczema - Testing of a Prevention-concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Allergy Research Center, Denmark (Other)
Collaborators: Arbejdsmiljøforskningsfonden (Unknown); Bispebjerg Hospital (Other); Frederiksberg University Hospital (Other); National Research Centre for the Working Environment, Denmark (Other Government); University of Osnabrueck (Other)
Responsible Party: Principal Investigator, Jojo Biel-Nielsen Dietz, Medical doctor, Ph.d.-student, National Allergy Research Center, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P-2019-650
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Occupational Contact Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Treatment in a hospital setting at Gentofte Hospital skin department with patient education, glove counselling, personal product screening by a chemistry engineer, extended allergy testing and the standard treatment of hand eczema.
  Interventions: Other: Treatment at the skin department at Gentofte Hospital
- Control group (No Intervention): Treatment as usual (at a dermatologist office).

INTERVENTIONS:
Other: Treatment at the skin department at Gentofte Hospital — Treatment in a hospital setting at Gentofte Hospital skin department
  Arms: Intervention group

SUMMARY:
Randomised controlled trial examining the effect of decreased waiting time for the first doctors' appointment, patient education, glove counselling and counselling at departments of social or occupational medicine on severity of hand eczema, quality of life, use of corticosteroids, and jobsituation 3-12 months after intervention in patients with suspected occupational contact dermatitis of the hands.

DETAILED DESCRIPTION:
Patients with suspected occupational hand eczema are recruited to the study on basis of their referral from general practitioner to dermatologist. Patients are randomised to either control or intervention group. The control group is treated and followed-up by the dermatologist they have been referred to, while the intervention group is treated and followed-up at Gentofte Hospital skin department with a maximum waiting time of 3 weeks. At the skin department at Gentofte Hospital, the patients in the intervention group receive patient education in prevention and treatment of hand eczema, glove counselling, personal product screening by a chemistry engineer, extended allergy testing and the standard treatment of hand eczema. Patients in both the control and intervention group are asked to fill out a questionnaire at 3, 6, 9 and 12 months after inclusion in the study. The questionnaire contains questions about quality of life, severity of hand exzema, jobsituation, use of healthcare service and use of medicine. Furthermore, prescriptions of medicine are registered in both control and intervention group at 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Referred from a general practitioner to a dermatologist
* Hand eczema within the last 3 months
* Suspicion that the hand eczema is work-related (either patient and/or doctors suspicion)

Exclusion Criteria:

* Does not read and write danish
* Severe psychiatric illness
* Pregnancy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Change in severity of handeczema assessed by the hand eczema severity index (HECSI) 0-360 points (0 best, 360 worst) | Change between baseline and 3 months
  The hand eczema severity index (HECSI)
Change in severity of handeczema assessed by the photographic guide for severity of handeczema | Change between baseline and 3 months
  Self-assessed photographic guide
Change in severity of handeczema assessed by the photographic guide for severity of handeczema | Change between baseline and 6 months
  Self-assessed photographic guide
Change in severity of handeczema assessed by the photographic guide for severity of handeczema | Change between baseline and 9 months
  Self-assessed photographic guide
Change in severity of handeczema assessed by the photographic guide for severity of handeczema | Change between baseline and 12 months
  Self-assessed photographic guide
Change in severity of handeczema assessed by a visual analog score 0-100 (0 best, 100 worst) | Change between baseline and 3 months
  Visual analog Score for severity of handeczema
Change in severity of handeczema assessed by a visual analog score 0-100 (0 best, 100 worst) | Change between baseline and 6 months
  Visual analog Score for severity of handeczema
Change in severity of handeczema assessed by a visual analog score 0-100 (0 best, 100 worst) | Change between baseline and 9 months
  Visual analog Score for severity of handeczema
Change in severity of handeczema assessed by a visual analog score 0-100 (0 best, 100 worst) | Change between baseline and 12 months
  Visual analog Score for severity of handeczema
Amount of corticosteroids prescribed within the last year | Baseline
  Amount of corticosteroids prescribed wihtin the last year
Amount of corticosteroids prescribed within the last 3 months | 3 months
  Amount of corticosteroids prescribed within the last 3 months
Amount of corticosteroids prescribed within the last 3 months | 6 months
  Amount of corticosteroids prescribed within the last 3 months
Amount of corticosteroids prescribed within the last 3 months | 9 months
  Amount of corticosteroids prescribed within the last 3 months
Amount of corticosteroids prescribed within the last 3 months | 12 months
  Amount of corticosteroids prescribed within the last 3 months
Health-Related Quality of Life assessed by Skindex-29, scale ranging from 0-100 points (higher score = higher impact of skin disease on quality of life) | Baseline
  Skindex-29
Health-Related Quality of Life assessed by Skindex-29, scale ranging from 0-100 points (higher score = higher impact of skin disease on quality of life) | 3 months
  Skindex-29
Health-Related Quality of Life assessed by Skindex-29, scale ranging from 0-100 points (higher score = higher impact of skin disease on quality of life) | 6 months
  Skindex-29
Health-Related Quality of Life assessed by Skindex-29, scale ranging from 0-100 points (higher score = higher impact of skin disease on quality of life) | 9 months
  Skindex-29
Health-Related Quality of Life assessed by Skindex-29, scale ranging from 0-100 points (higher score = higher impact of skin disease on quality of life) | 12 months
  Skindex-29
Health-Related Quality of Life assessed by "European Quality of Life - 5 Dimensions" (EQ-5D) | Baseline
  "European Quality of Life - 5 Dimensions" (EQ-5D)
Health-Related Quality of Life assessed by "European Quality of Life - 5 Dimensions" (EQ-5D) | 3 months
  "European Quality of Life - 5 Dimensions" (EQ-5D)
Health-Related Quality of Life assessed by "European Quality of Life - 5 Dimensions" (EQ-5D) | 6 months
  "European Quality of Life - 5 Dimensions" (EQ-5D)
Health-Related Quality of Life assessed by "European Quality of Life - 5 Dimensions" (EQ-5D) | 9 months
  "European Quality of Life - 5 Dimensions" (EQ-5D)
Health-Related Quality of Life assessed by "European Quality of Life - 5 Dimensions" (EQ-5D) | 12 months
  "European Quality of Life - 5 Dimensions" (EQ-5D)
Health-Related Quality of Life assessed by Dermatology life quality index (DLQI) 0-30 (higher score = higher impact of skin disease on quality of life) | Baseline
  Dermatology life quality index (DLQI)
Health-Related Quality of Life assessed by Dermatology life quality index (DLQI) 0-30 (higher score = higher impact of skin disease on quality of life) | 3 months
  Dermatology life quality index (DLQI)
Health-Related Quality of Life assessed by Dermatology life quality index (DLQI) 0-30 (higher score = higher impact of skin disease on quality of life) | 6 months
  Dermatology life quality index (DLQI)
Health-Related Quality of Life assessed by Dermatology life quality index (DLQI) 0-30 (higher score = higher impact of skin disease on quality of life) | 9 months
  Dermatology life quality index (DLQI)
Health-Related Quality of Life assessed by Dermatology life quality index (DLQI) 0-30 (higher score = higher impact of skin disease on quality of life) | 12 months
  Dermatology life quality index (DLQI)
Number of participants with loss of job within the last year | Baseline
  Self-repported loss of job wihtin the last year
Number of participants with loss of job within the last 3 months | Baseline
  Self-repported loss of job within the last 3 months
Number of participants with loss of job within the last 3 months | 3 months
  Self-repported loss of job within the last 3 months
Number of participants with loss of job within the last 3 months | 6 months
  Self-repported loss of job within the last 3 months
Number of participants with loss of job within the last 3 months | 9 months
  Self-repported loss of job within the last 3 months
Number of participants with loss of job within the last 3 months | 12 months
  Self-repported loss of job within the last 3 months
Amount of sick leave within the last year | Baseline
  Self-repported amount of sick leave within the last year
Amount of sick leave within the last 3 months | 3 months
  Self-repported amount of sick leave within the last 3 months
Amount of sick leave within the last 3 months | 6 months
  Self-repported amount of sick leave within the last 3 months
Amount of sick leave within the last 3 months | 9 months
  Self-repported amount of sick leave within the last 3 months
Amount of sick leave within the last 3 months | 12 months
  Self-repported amount of sick leave within the last 3 months
Number of participants with change of occupation due to occupational contact dermatitis within the last year | Baseline
  Change of occupation due to occupational contact dermatitis within the last year
Number of participants with change of occupation due to occupational contact dermatitis within the last 3 months | 3 months
  Change of occupation due to occupational contact dermatitis within the last 3 months
Number of participants with change of occupation due to occupational contact dermatitis within the last 3 months | 6 months
  Change of occupation due to occupational contact dermatitis within the last 3 months
Number of participants with change of occupation due to occupational contact dermatitis within the last 3 months | 9 months
  Change of occupation due to occupational contact dermatitis within the last 3 months
Number of participants with change of occupation due to occupational contact dermatitis within the last 3 months | 12 months
  Change of occupation due to occupational contact dermatitis within the last 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne D Johansen, Professor, Study Director — National Allergy Research Center
Locations (1):
- Gentofte Hospital, Skin department, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No